CLINICAL TRIAL: NCT05054348
Title: A Phase 1b, Open-Label, Dose-Escalation, Dose-Expansion, and Dose-Randomization Study of IO 108 as Monotherapy and in Combination With Either Pembrolizumab or Cemiplimab in Adult Patients With Advanced Solid Tumors
Brief Title: First-in-human Study of IO-108 as Single Agent and in Combination With a PD-1 Immune Check Point Inhibitor in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Immune-Onc Therapeutics (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IO-108-CL-001
Record Dates: First submitted 2021-08-30; First posted 2021-09-23 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-03

CONDITIONS: Solid Tumor, Adult
Keywords: IO-108

STUDY DESIGN:
Intervention Model Description: Dose escalation, dose expansion and dose randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- IO-108 Monotherapy (Experimental): Treatment of patients with advanced solid tumors with IO-108 monotherapy
  Interventions: Biological: IO-108
- IO-108 + pembrolizumab combination therapy (Experimental): Treatment of patients with advanced solid tumors with IO-108 in combination with a fixed dose of pembrolizumab
  Interventions: Biological: IO-108 + pembrolizumab combination therapy
- IO-108 + cemiplimab combination therapy (Experimental): Treatment of patients with advanced solid tumors with IO-108 in combination with a fixed dose of cemiplimab
  Interventions: Biological: IO-108 + cemiplimab combination therapy

INTERVENTIONS:
Biological: IO-108 — IO-108 given as monotherapy
  Arms: IO-108 Monotherapy
Biological: IO-108 + pembrolizumab combination therapy — IO-108 and fixed dose pembrolizumab combination therapy
  Other Names: IO-108 + Keytruda combination therapy
  Arms: IO-108 + pembrolizumab combination therapy
Biological: IO-108 + cemiplimab combination therapy — IO-108 and fixed dose cemiplimab combination therapy
  Other Names: IO-108 + Libtayo combination therapy
  Arms: IO-108 + cemiplimab combination therapy

SUMMARY:
The goal of the clinical trial is to learn about safety, tolerability and preliminary efficacy of IO-108 as monotherapy or in combination with a PD-1 inhibitor in patients with advanced, metastatic solid tumors, and to find a dose of IO-108 that is safe and efficacious to be tested in patients with various solid tumors.

DETAILED DESCRIPTION:
In the Part 1 Dose Escalation, safety and tolerability of varying doses of IO-108 as monotherapy or in combination with pembrolizumab will be studied, in order to determine a proposed RP2D. In Part 2 Dose Expansion, patients with various types of solid tumors will be dosed with either IO-108 alone or in combination with either pembrolizumab or cemiplimab in order to study safety, tolerability and preliminary efficacy of IO-108 monotherapy and combination with a PD-1 inhibitor. In Part 3, a tumor type that has been studied in the Dose Expansion will be selected and patients will be randomized into 2 doses of IO-108 in order to explore safety, toxicity, efficacy relationship with exposure, in order to explore different doses of IO-108 that is safe and efficacious. Safety, PK, PD biomarkers and efficacy will be studied.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be ≥18.
2. Has any histologically- or cytologically confirmed advanced/metastatic solid tumor by pathology report and has received, has been intolerant to, or has been ineligible for standard systemic therapy known to confer clinical benefit. Solid tumors of any type are eligible for enrollment. Patients with asymptomatic central nervous system (CNS) disease may be enrolled.
3. Patient has measurable disease by Response Evaluation in Solid Tumors version 1.1 (RECIST 1.1) as assessed by local site.
4. Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
5. Patients must have adequate hepatic function and renal function.

Exclusion Criteria:

1. Patients who previously received a monoclonal antibody therapy targeting LILRB2/ Immunoglobulin-Like Transcript 4 (ILT4) (including IO-108).
2. Patients who received a biologic systemic anti-cancer therapy <4 weeks or 5 half-lives prior to their first day of study drug administration, or a small molecule systemic anti-cancer therapy or definitive radiotherapy <2 weeks or 5 half-lives prior to their first day of study drug administration or have not recovered to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0 Grade 1 or better from any adverse events (AEs) that were due to prior cancer therapeutics. Palliative radiation is allowed within 2 weeks of the first day of study drug administration.
3. Requires systemic corticosteroids at a dose of >10 mg prednisone or the dose equivalent to other systemic corticosteroid.
4. History of radiation pneumonitis, non-infectious pneumonitis or interstitial lung disease.
5. Symptomatic CNS spread of tumor.
6. History of Grade > 3 immune-related AEs with any prior immunotherapy.
7. Patients with uncontrolled, active infection.
8. Patients with known hypersensitivity to any of the components of the IO-108 formulation or pembrolizumab.
9. Active known malignancy with the exception of any of the following:

   1. Adequately treated basal cell carcinoma, squamous cell carcinoma of the skin, or in situ cervical cancer;
   2. Low-risk prostate cancer for which observation or hormonal therapy only is indicated;
   3. Any other malignancy treated with curative intent with the last treatment completed ≥6 months before study initiation (with the exception of hormonal therapies when indicated).
10. Patients with New York Heart Association (NYHA) Class III or IV congestive heart failure (CHF) or left ventricular ejection fraction (LVEF) <40% by echocardiogram (ECHO) or multi-gated acquisition (MUGA) scan ≤28 days prior to Cycle 1 Day 1 (C1D1).
11. Any of the following in the previous 6 months: myocardial infarction, congenital long QT syndrome, Torsades de pointes, clinically significant arrhythmias (including sustained ventricular tachyarrhythmia and ventricular fibrillation), and left anterior hemiblock (bifascicular block), unstable angina, coronary/peripheral artery bypass graft, symptomatic CHF (NYHA class III or IV), cerebrovascular accident, transient ischemic attack, or pulmonary embolism. Patients with asymptomatic right bundle branch block or controlled atrial fibrillation are allowed.
12. Ongoing cardiac dysrhythmias of Grade 2 or higher per NCI CTCAE, Version 5.0.
13. Known active bacterial, viral, and/or fungal infection including hepatitis B (HBV), hepatitis C, human immunodeficiency virus (HIV), severe acute respiratory syndrome coronavirus 2 (SARS-COV-2) or acquired immunodeficiency syndrome (AIDS)-related illness.
14. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent and serious adverse events in patients treated with IO-108 and IO-108+pembrolizumab | From first dose of IO-108 until the end of treatment which is up to 2 years from the first treatment date or disease progression whichever is earlier
  safety and tolerability as measured by the incidence of treatment-emergent adverse events and serious adverse events
Determine MTD (maximum tolerated dose) through assessment of dose-limiting toxicities (DLT) | From the first dose of IO-108 until 21 days post-treatment
  MTD will be determined through observation of pre-determined DLTs in each dose cohort
Assess safety and tolerability of the IO-108 RP2D as monotherapy or in combination with either pembrolizumab or cemiplimab in patients with solid tumors | From the first dose of IO-108 until the end of treatment which is up to 2 years from the first treatment or disease progression, whicheer is earlier
  safety and tolerability as measured by the incidence of treatment-emergent adverse events and discontinuation due to TEAEs

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of IO-108 | From the first dose of IO-108 until day 15 post-treatment
  Characterize the Cmax of IO-108 by successive sampling of blood at pre-specified time points
Steady state concentration of IO-108 | From the second dose of IO-108 until the last treatment which is up to 2 years from the first treatment date
  Characterize steady state concentration of IO-108 by successive sampling of blood at pre-specified time points
Immunogenicity of IO-108 and IO-108+pembrolizumab | From the first dose until 30 days after the last treatment
  Determine the incidence/titer of anti-drug antibodies (ADAs) against IO-108 and pembrolizumab (in combination treatment)
Anti-tumor activity of IO-108 and IO-108+pembrolizumab | From the date of first treatment until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to estimated period of 48 months
  Determine preliminary rates of response after treatment with IO-108
Determine disease control rates of IO-108 as monotherapy or in combination with either pembrolizumab or cemiplimab | From the first dose of IO-108 until the last treatment which is up to 2 years from the first treatment or disease progression whichever is earlier
  Disease control rate is defined as the percentage of patients with complete response, partial response or stable disease maintained for at least 3 months

OTHER OUTCOMES:
Receptor occupancy of IO-108 in IO-108 monotherapy and IO-108+pembrolizumab | From the first dose of IO-108 till 21 days after
  To assess target engagement via determining Leukocyte Immunoglobulin-Like Receptor subfamily B2 (LILRB2) occupancy by IO-108 in peripheral blood myeloid cells, as expressed by % of target receptor engagement

CONTACTS AND LOCATIONS:
Overall Officials: Wen Hong Lin, MD, Study Director — Immune-Onc Therapeutics
Locations (24):
- United States (24):
  - Arizona Oncology Associates, PC-HOPE (140) (USOR SITE), Tucson, Arizona
  - Beverly HIlls Cancer Center (129), Beverly Hills, California
  - Rocky Mountain Cancer Centers, LLP (141) (USOR SITE), Lone Tree, Colorado
  - University of Florida (125), Gainesville, Florida
  - Florida Cancer Specialists (134), Lake Mary, Florida
  - Memorial Cancer Institute (146), Pembroke Pines, Florida
  - Florida Cancer Specialists & Research Institute (103), Sarasota, Florida
  - Hematology Oncology (136), Stuart, Florida
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center (123), Indianapolis, Indiana
  - Maryland Oncology Hematology, PA (145) (USOR SITE), Columbia, Maryland
  - Karmanos Cancer Institute (126), Detroit, Michigan
  - St. Vincent - Frontier Cancer Center (135), Billings, Montana
  - NYU Langone Health (131), New York, New York
  - Carolina BioOncology (102), Huntsville, North Carolina
  - Gabrail Cancer Center (128), Canton, Ohio
  - Oncology Hematology Care Clinical Trials, LLC (144) (USOR SITE), Cincinnati, Ohio
  - Providence Cancer Institute (104), Portland, Oregon
  - UPMC Hillman Cancer Center (105), Pittsburgh, Pennsylvania
  - Texas Oncology - Austin (142) (USOR SITE), Austin, Texas
  - Texas Oncology - Baylor Charles A. (143) (USOR SITE), Dallas, Texas
  - MD Anderson Cancer Center (101), Houston, Texas
  - Oncology Consultants, P.A. (138), Houston, Texas
  - NEXT Oncology-Virginia (121), Fairfax, Virginia
  - Swedish Cancer Institute (147), Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Taylor MH, Naing A, Powderly J, Woodard P, Chung L, Lin WH, Tian H, Siemers N, Xiang H, Deng R, Hong K, Valencia D, Huang T, Zhu Y, Liao XC, Schebye XM, Patel MR. Phase I dose escalation study of IO-108, an anti-LILRB2 antibody, in patients with advanced solid tumors. J Immunother Cancer. 2024 Nov 20;12(11):e010006. doi: 10.1136/jitc-2024-010006. PMID 39567210